CLINICAL TRIAL: NCT06499038
Title: Migration Analysis of a Hybrid Hip Replacement Evaluating Stem and Ancillary Acetabular Screw Fixation-A Randomized Controlled CT-RSA Trial
Brief Title: The Ace Avanteon Study - A Randomized Controled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Helse Møre og Romsdal HF (Other Government)
Collaborators: St. Olavs Hospital (Other); JRI Orthopaedics Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 536698
Record Dates: First submitted 2024-06-03; First posted 2024-07-12 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Hip Osteoarthritis
Keywords: , Total Hip Arthroplasty,; Total Hip Replacement; CT-RSA; CTMA; Migration study
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Intervention Model Description: Randomized controled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ancillary screw group (Experimental): Patients with ancillary screw fixation acetabular component
  Interventions: Procedure: Total Hip Arthroplasty
- Without ancillary screws group (Active Comparator): No ancillary screws in acetabular component
  Interventions: Procedure: Total Hip Arthroplasty

INTERVENTIONS:
Procedure: Total Hip Arthroplasty — Surgery for total hip replacement
  Other Names: ACE cup and Avanteon Stem

SUMMARY:
The goal of this randomized controled trial is to compare if using of ancillary screws yields equal results as no use of ancillary screws in the ACE acetabulum cup of a total hip arthroplasty. Further, the migration of the Avanteon stem over time will be assessed. Patients included are patients with hip osteoarthritis from 65-80 years old. The purpose of this study is to compare implant migration and early fixation of a hybrid hip replacement combining the uncemented ACE acetabular component and the cemented Avanteon femoral stem, by using CT based Radiostereometric Analysis, a new innovative method for evaluating implant migration. Our study may predict the long term survival of the implants used.

Participants will go through total hip arthroplasty, and be followed by CT-RSA, plain x-rays and patients reported outcome measures.

DETAILED DESCRIPTION:
Hip and knee osteoarthritis OA is one of the leading causes of disability worldwide. The lifetime risk of developing hip OA is estimated to be 25%, in people who reach the age of 85. Total hip replacement THR is considered to be a safe and reliable surgical treatment for end stage hip OA and was described as "Surgery of the century". One of the challenges in hip replacement surgery is to ensure the longevity and durability of the implants used. New implants are designed to improve the primary stability and long-term survival of the implant. Early failure of implants and the need for revision surgery, is a major concern. Revision hip replacement surgery is a surgical procedure with high rates of postoperative complications and overall re-revision rate of 15,8% within 1 year. In the Norwegian arthroplasty register 10 year failure rate of hip revision prostheses is 26%. Thus, the longevity and durability of implants is a continuous challenge in which the ultimate goal is to develop well-functioning implants which will last a lifetime.

The purpose of this study is to compare implant migration and early fixation of a hybrid hip replacement combining the uncemented ACE acetabular component and the cemented Avanteon femoral stem, by using CT based Radiostereometric Analysis, a new innovative method for evaluating implant migration. Our study may predict the long term survival of the implants used. This will be the first ever CT-RSA study in Norway and one of the first world-wide, evaluating hip implants.

Radiostereometric analysis RSA is a method used to measure implant migration and micromotion after joint replacement surgery, with high precision and accuracy. It is considered the gold standard for to assess migration in orthopedic implants. Early implant migration predicts later loosening, and failure of the implant. Subsidence of the femoral stem of more than 1.2 mm at 24m months is predictive of revision. Proximal migration of the acetabular component of up to 0.2mm is considered acceptable, 0.2-1mm is considered at risk, and above 1mm is unacceptable. RSA is thereby used as an early measure of longevity and durability of new implants. However, RSA is an expensive and time consuming procedure. It requires special equipment such as RSA cages, software, and special x-ray setup. It also requires specially trained personnel to do the examination. Loss of data due to occlusion of tantalum beads from metallic implants, is unavoidable in RSA. Over the last years CT-RSA has evolved to overcome some of the challenges of RSA. CT-RSA has been validated to have similar or even higher precision and accuracy than RSA in both hip and knee implant analysis.By using CT-RSA we can evaluate implant migration without the need for implant or bone markers, by using bone surface anatomy. One of the authors (FDØ) has recently shown that a vast decrease of effective radiation doses of CT-RSA in total knee arthroplasty yields equal precision in a cadaver study (publication in press). We assume this applies to CT-RSA of the hip as well. We therefore would like to perform a study on ultra low dose CT-RSA of hip implants, to evaluate the precision. This could have a major impact for future CT-RSA studies of the hip, since we potentially could reduce the effective radiation dose.

Previous cadaveric studies have shown that screw fixation increases initial stability of acetabular components. In long term, press-fit screwless fixation achieve sufficient stability.The use of augmented screw fixation may increase the risk of particle debris and osteolysis around the acetabular component. The use of ancillary screw fixation may thereby increase the risk of loosening, and need for major revision surgery. There is also a risk for iatrogenic damage to nearby vessels and pelvic organs, due to screw misplacement.

The Avanteon JRI is a highly polished double tapered femoral stem, designed by force-closed principles. The stem is intended to subside gradually in the cement mantle over time. Highly polished femoral stems have shown excellent results, and lower revision rates compared to shape-closed design stems. New implants are developed to increase early fixation and long term survival, to avoid the need for revision surgery.

In the field of orthopedic surgery, our study may predict the long term survival of the implants used, and thereby contributing to the goal of life-long lasting implants. This will also contribute to lower the need for revision surgery, avoiding the risk of major complications for our patients. The economic impact off revision surgery is of great concern for both the patient and the society, and avoiding the need for revision arthroplasty is of economic importance.

Research questions and goals In our study we will evaluate the migration of the Avanteon femoral stem using CT-RSA, to predict long-term survival. We will also evaluate the role of ancillary screw fixation of the new ACE acetabular component by using CT-RSA, to see if ancillary screw fixation increases stability of the implant. By using a patient attached accelerometer-based activity monitor ActivePAL, we can measure patient activity to see if the screw fixation has any effect on activity levels.

Hypotheses; Article 1

* H0-hypothesis; subsidence of the Avanteon femoral stem is less than 1.2mm at 24 months
* H1-hypothesis; subsidence of the Avanteon femoral stem is more than 1.2mm at 24 months

Article 2

* H0-hypothesis; ancillary screw fixation of the ACE acetabular component does not increase stability of the implant
* H1-hypothesis; ancillary screw fixation of the ACE acetabular component increases stability of the implant

Article 3

* H0-hypothesis; ancillary screw fixation of the ACE acetabular component does not increase patient activity
* H1-hypothesis; ancillary screw fixation of the ACE acetabular component increases patient activity

Article 4

* H0-hypothesis; reducing the effective radiation dose does not reduce the precision of CT-RSA of hip implants
* H1-hypothesis; reducing the effective radiation dose reduce the precision of CT-RSA of hip implants

Short term goals;

* Demonstrating the stability and migration of the Avanteon femoral stem
* Evaluate the stability and migration of the ACE acetabular component with and without ancillary screw fixation
* Demonstrate the clinical efficacy and safety of the ACE acetabular component and Avanteon femoral stem
* Demonstrate the effect of acetabular screw fixation on patient activity levels in the postoperative period Demonstrate the precision of ultra low dose CT-RSA Long term goals;
* Contributing to the development of longer lasting hip replacement implants
* Evaluate the increase in activity levels after hip replacement surgery

Results expected to be achieved during the project period;

* Establishing the new innovative CT-RSA as a method for hip implant migration analysis in Norway
* Develop recommendation for the routine use of ancillary screw fixation of acetabular components

This is a single blinded randomized controlled trial. Eligible patients referred will be evaluated for inclusion consecutively from the outpatient clinic of the research department at Kristiansund hospital.

ELIGIBILITY:
Inclusion Criteria:

* • Patients with primary hip osteoarthritis between the age of 65 and 80 years at time of surgery

  * Patients requiring primary total hip replacement
  * Patients who understand the conditions of the study, are willing to, and able to comply with the postoperative scheduled clinical and radiographic evaluations

Exclusion Criteria:

* • Patients who are unable to provide informed consent

  * Patients who require revision hip arthroplasty
  * Patients who have had a previous osteotomy or osteosynthesis of the femur or acetabulum
  * Patients with metabolic bone disease, other than osteoporosis
  * Patients with inflammatory arthritis
  * Obese patients where obesity is severe enough to affect the patient's ability to perform activities of daily living (BMI > 40)
  * Patients with active or suspected infection
  * Patients with malignancy
  * Patients unable to cooperate caused by language or psychosocial conditions

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-08-25 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Translation | 2 years
  Proximal Y migration acetabular cup measured by CT-RSA

SECONDARY OUTCOMES:
Rotation | 2 years
  Rotation XYZ measured by CT-RSA
Migration | 2 years
  Anterior and axial XZ migration acetabular cup measured by CT-RSA
MTPM | 2 years
  MTPM of acetabular cup
Stem Tr | 2 years
  Subsidence of stem
XZ translation of Avanteon stem | 2 years
  Migration
XYZ rotation | 2 years
  Rotation of stem in 3 dimensions

OTHER OUTCOMES:
Difference precision | 3 months
  Precision CT-RSA measured by double investigations at 2 different dose levels
PROMs | 2 years
  Patient reported outcome measures like EQ-5D-5L, OHS, VAS, FJS and HOOS

CONTACTS AND LOCATIONS:
Overall Officials: Frank-David Øhrn, MD, PhD, Study Chair — Møre og Romsdal Hospital Trust; Mathias Brevik, MD, Principal Investigator — Møre og Romsdal Hospital Trust; Otto Schnell Husby, Professor, Study Director — Norwegian University of Science and Technology; Kirsti Sevaldsen, MD, PHD, Study Chair — Møre og Romsdal Hospital Trust
Locations (1):
- Kristiansund Hospital, Møre and Romsdal Hospital Trust, Kristiansund, Møre and Romsdal, Norway

IPD SHARING:
Plan to Share IPD: Yes
Upon request with proper reasons, we will share data with other researchers including CT-RSA data and PROMs. This will of course be performed within the laws of Norway and totally anonymized.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: From 3 years from now and as long as the data is stored.
Access Criteria: Proper request to the corresponding author.

REFERENCES:
- [Background] Murphy LB, Helmick CG, Schwartz TA, Renner JB, Tudor G, Koch GG, Dragomir AD, Kalsbeek WD, Luta G, Jordan JM. One in four people may develop symptomatic hip osteoarthritis in his or her lifetime. Osteoarthritis Cartilage. 2010 Nov;18(11):1372-9. doi: 10.1016/j.joca.2010.08.005. Epub 2010 Aug 14. PMID 20713163
- [Background] Learmonth ID, Young C, Rorabeck C. The operation of the century: total hip replacement. Lancet. 2007 Oct 27;370(9597):1508-19. doi: 10.1016/S0140-6736(07)60457-7. PMID 17964352
- [Background] Badarudeen S, Shu AC, Ong KL, Baykal D, Lau E, Malkani AL. Complications After Revision Total Hip Arthroplasty in the Medicare Population. J Arthroplasty. 2017 Jun;32(6):1954-1958. doi: 10.1016/j.arth.2017.01.037. Epub 2017 Feb 1. PMID 28236550
- [Background] Lie SA, Havelin LI, Furnes ON, Engesaeter LB, Vollset SE. Failure rates for 4762 revision total hip arthroplasties in the Norwegian Arthroplasty Register. J Bone Joint Surg Br. 2004 May;86(4):504-9. PMID 15174543
- [Background] Selvik G. Roentgen stereophotogrammetry. A method for the study of the kinematics of the skeletal system. Acta Orthop Scand Suppl. 1989;232:1-51. PMID 2686344
- [Background] Valstar ER, Gill R, Ryd L, Flivik G, Borlin N, Karrholm J. Guidelines for standardization of radiostereometry (RSA) of implants. Acta Orthop. 2005 Aug;76(4):563-72. doi: 10.1080/17453670510041574. PMID 16195075
- [Background] Karrholm J, Borssen B, Lowenhielm G, Snorrason F. Does early micromotion of femoral stem prostheses matter? 4-7-year stereoradiographic follow-up of 84 cemented prostheses. J Bone Joint Surg Br. 1994 Nov;76(6):912-7. PMID 7983118
- [Background] Ryd L, Albrektsson BE, Carlsson L, Dansgard F, Herberts P, Lindstrand A, Regner L, Toksvig-Larsen S. Roentgen stereophotogrammetric analysis as a predictor of mechanical loosening of knee prostheses. J Bone Joint Surg Br. 1995 May;77(3):377-83. PMID 7744919
- [Background] Pijls BG, Nieuwenhuijse MJ, Fiocco M, Plevier JW, Middeldorp S, Nelissen RG, Valstar ER. Early proximal migration of cups is associated with late revision in THA: a systematic review and meta-analysis of 26 RSA studies and 49 survivalstudies. Acta Orthop. 2012 Dec;83(6):583-91. doi: 10.3109/17453674.2012.745353. Epub 2012 Nov 5. PMID 23126575
- [Background] Broden C, Sandberg O, Olivecrona H, Emery R, Skoldenberg O. Precision of CT-based micromotion analysis is comparable to radiostereometry for early migration measurements in cemented acetabular cups. Acta Orthop. 2021 Aug;92(4):419-423. doi: 10.1080/17453674.2021.1906082. Epub 2021 Apr 6. PMID 33821746
- [Background] Otten V, Maguire GQ Jr, Noz ME, Zeleznik MP, Nilsson KG, Olivecrona H. Are CT Scans a Satisfactory Substitute for the Follow-Up of RSA Migration Studies of Uncemented Cups? A Comparison of RSA Double Examinations and CT Datasets of 46 Total Hip Arthroplasties. Biomed Res Int. 2017;2017:3681458. doi: 10.1155/2017/3681458. Epub 2017 Jan 24. PMID 28243598
- [Background] Engseth LHW, Schulz A, Pripp AH, Rohrl SMH, Ohrn FD. CT-based migration analysis is more precise than radiostereometric analysis for tibial implants: a phantom study on a porcine cadaver. Acta Orthop. 2023 Apr 27;94:207-214. doi: 10.2340/17453674.2023.12306. PMID 37114404
- [Background] Burkhart TA, Khadem M, Wood TJ, Dunning CE, Degen R, Lanting BA. Comparison of trans-cortical and cancellous screws to press fit for acetabular shell fixation in total hip arthroplasty: A cadaveric study. Clin Biomech (Bristol). 2019 Oct;69:34-38. doi: 10.1016/j.clinbiomech.2019.06.017. Epub 2019 Jun 28. PMID 31295668
- [Background] Otten VT, Crnalic S, Rohrl SM, Nivbrant B, Nilsson KG. Stability of Uncemented Cups - Long-Term Effect of Screws, Pegs and HA Coating: A 14-Year RSA Follow-Up of Total Hip Arthroplasty. J Arthroplasty. 2016 Jan;31(1):156-61. doi: 10.1016/j.arth.2015.07.012. Epub 2015 Jul 11. PMID 26260783
- [Background] Brodt S, Bischoff K, Schulze M, Nowack D, Roth A, Matziolis G. The use of acetabular screws in total hip arthroplasty and its influence on wear and periacetabular osteolysis in the long-term follow-up. Int Orthop. 2022 Apr;46(4):717-722. doi: 10.1007/s00264-021-05219-7. Epub 2021 Sep 28. PMID 34581866
- [Background] Alshameeri Z, Bajekal R, Varty K, Khanduja V. Iatrogenic vascular injuries during arthroplasty of the hip. Bone Joint J. 2015 Nov;97-B(11):1447-55. doi: 10.1302/0301-620X.97B11.35241. PMID 26530643
- [Background] Ayob KA, Merican AM, Sulaiman SH, Hariz Ramli AR. The tale of two vessels, vascular complications following a breach of the pelvic inner table due to acetabular screws: a report of two cases. Jt Dis Relat Surg. 2021;32(1):239-244. doi: 10.5606/ehc.2021.77862. PMID 33463444
- [Background] Kinmont JC. Penetrating bladder injury caused by a medially placed acetabular screw. J South Orthop Assoc. 1999 Summer;8(2):98-100. PMID 10472827
- [Background] Keeling P, Howell JR, Kassam AM, Sathu A, Timperley AJ, Hubble MJW, Wilson MJ, Whitehouse SL. Long-Term Survival of the Cemented Exeter Universal Stem in Patients 50 Years and Younger: An Update on 130 Hips. J Arthroplasty. 2020 Apr;35(4):1042-1047. doi: 10.1016/j.arth.2019.11.009. Epub 2019 Nov 14. PMID 31882346
- [Background] Ling RS, Charity J, Lee AJ, Whitehouse SL, Timperley AJ, Gie GA. The long-term results of the original Exeter polished cemented femoral component: a follow-up report. J Arthroplasty. 2009 Jun;24(4):511-7. doi: 10.1016/j.arth.2009.02.002. Epub 2009 Mar 17. PMID 19282139
- [Background] Mahon J, McCarthy CJ, Sheridan GA, Cashman JP, O'Byrne JM, Kenny P. Outcomes of the Exeter V40 cemented femoral stem at a minimum of ten years in a non-designer centre. Bone Jt Open. 2020 Dec 7;1(12):743-748. doi: 10.1302/2633-1462.112.BJO-2020-0163.R1. PMID 33367281
- [Background] Ryan CG, Grant PM, Tigbe WW, Granat MH. The validity and reliability of a novel activity monitor as a measure of walking. Br J Sports Med. 2006 Sep;40(9):779-84. doi: 10.1136/bjsm.2006.027276. Epub 2006 Jul 6. PMID 16825270
- [Background] Taraldsen K, Askim T, Sletvold O, Einarsen EK, Bjastad KG, Indredavik B, Helbostad JL. Evaluation of a body-worn sensor system to measure physical activity in older people with impaired function. Phys Ther. 2011 Feb;91(2):277-85. doi: 10.2522/ptj.20100159. Epub 2011 Jan 6. PMID 21212377
- [Background] Moher D, Hopewell S, Schulz KF, Montori V, Gotzsche PC, Devereaux PJ, Elbourne D, Egger M, Altman DG. CONSORT 2010 explanation and elaboration: updated guidelines for reporting parallel group randomised trials. BMJ. 2010 Mar 23;340:c869. doi: 10.1136/bmj.c869. No abstract available. PMID 20332511
- [Background] Derbyshire B, Prescott RJ, Porter ML. Notes on the use and interpretation of radiostereometric analysis. Acta Orthop. 2009 Feb;80(1):124-30. doi: 10.1080/17453670902807474. PMID 19234894
- [Background] Engdal M, Foss OA, Taraldsen K, Husby VS, Winther SB. Daily Physical Activity in Total Hip Arthroplasty Patients Undergoing Different Surgical Approaches: A Cohort Study. Am J Phys Med Rehabil. 2017 Jul;96(7):473-478. doi: 10.1097/PHM.0000000000000657. PMID 28628534
- [Background] Husby OS, Haugan K, Benum P, Foss OA. A prospective randomised radiostereometric analysis trial of SmartSet HV and Palacos R bone cements in primary total hip arthroplasty. J Orthop Traumatol. 2010 Mar;11(1):29-35. doi: 10.1007/s10195-010-0087-x. Epub 2010 Mar 3. PMID 20198403
- [Background] Sevaldsen K, S Husby O, B Lian O, S Husby V. Does the line-to-line cementing technique of the femoral stem create an adequate cement mantle? Hip Int. 2021 Sep;31(5):618-623. doi: 10.1177/1120700020934368. Epub 2020 Jun 18. PMID 32551930
- [Background] Sevaldsen K, Schnell Husby O, Lian OB, Farran KM, Schnell Husby V. Is the French Paradox cementing philosophy superior to the standard cementing? A randomized controlled radiostereometric trial and comparative analysis. Bone Joint J. 2022 Jan;104-B(1):19-26. doi: 10.1302/0301-620X.104B1.BJJ-2021-0325.R2. PMID 34969272
- [Background] Ohrn FD, Lian OB, Tsukanaka M, Rohrl SM. Early migration of a medially stabilized total knee arthroplasty : a radiostereometric analysis study up to two years. Bone Jt Open. 2021 Sep;2(9):737-744. doi: 10.1302/2633-1462.29.BJO-2021-0115.R1. PMID 34493056
- [Background] Ohrn FD, Van Leeuwen J, Tsukanaka M, Rohrl SM. A 2-year RSA study of the Vanguard CR total knee system: A randomized controlled trial comparing patient-specific positioning guides with conventional technique. Acta Orthop. 2018 Aug;89(4):418-424. doi: 10.1080/17453674.2018.1470866. Epub 2018 May 9. PMID 29739264
- [Background] Scheerlinck T, Polfliet M, Deklerck R, Van Gompel G, Buls N, Vandemeulebroucke J. Development and validation of an automated and marker-free CT-based spatial analysis method (CTSA) for assessment of femoral hip implant migration: In vitro accuracy and precision comparable to that of radiostereometric analysis (RSA). Acta Orthop. 2016;87(2):139-45. doi: 10.3109/17453674.2015.1123569. Epub 2015 Dec 3. PMID 26634843
- [Background] Boettner F, Sculco P, Lipman J, Renner L, Faschingbauer M. A novel method to measure femoral component migration by computed tomography: a cadaver study. Arch Orthop Trauma Surg. 2016 Jun;136(6):857-63. doi: 10.1007/s00402-016-2442-8. Epub 2016 Mar 16. PMID 26983723
- See also: ICMJE recommendations — http://www.icmje.org/